CLINICAL TRIAL: NCT01792141
Title: The Use of Fluorescein-Indocyanine Green Angiography in Patients With Diabetic Macular Edema to Identify Areas of Increased Leakage and Provide Targeted Focal Laser Treatment.
Brief Title: Use of Diagnostic Dye to Identify Areas of Leakeage,in the Retina, Prior to Receiving Focal Laser Treatment
Status: Completed | Type: Observational
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: RIH 1010
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of Indocyanine green diagnostic dye will identify areas of vascular leakage which will provide more effective laser treatment by targeting these specific areas.

DETAILED DESCRIPTION:
The Early Treatment of Diabetic Retinopathy Study showed that early treatment of Clinically Significant Macular Edema (CSME) with focal and grid laser preserved vision in diabetic patients. Indocyanine Green angiography, which was not available at the time of the Early Treatment Diabetic Retinopathy Study (ETDRS), is now standard-of-care for diagnostic evaluation of the choroidal circulation and is routinely done in combination with Fluorescein angiography for a more complete visualization of retinal pathology. Simultaneous examination of both retinal and choroidal circulation allows for identification of microaneurysms that are hyperfluorescent both on Fluorescein angiography and Indocyanine green angiography. Such microaneurysms are sites of increased vascular leakage and represent a means for providing more effective laser treatment by targeting these areas directly with focal laser.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Clinically Significant Macular Edema
* Microaneurysms hyperfluorescent

Exclusion Criteria:

* Increase intraocular pressure
* Intraocular inflammation
* Retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Clinically Significant Macular Edema
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary objective is to assess the effectiveness of FA-ICG guided focal laser therapy for the treatment CSME by means of serial FA-1CGs before and every 3 months after treatment. | 3 months
  Visual Acuity will be measured by using the Early Treatment Diabetic Retinopathy Study. (ETDRS) Macular volume will be measured by Optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Bennett, MD, Principal Investigator — Retina Institute of Hawaii
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States